CLINICAL TRIAL: NCT00323336
Title: Salivary Markers of Bone Turnover Compared to Urine and Blood
Brief Title: Markers of Bone Turnover in Saliva and How This Compares to Urine and Blood
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Other Study IDs: 77-05
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Last update posted 2010-01-25 (Estimated); Status verified 2010-01

CONDITIONS: Bone Turnover Markers; Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Study is being done to determine if it is possible to use saliva to measure bone specific proteins and predict bone turnover which could be used in the treatment of osteoporosis.

DETAILED DESCRIPTION:
Prevention and treatment of osteoporosis require sensitive and specific assays of bone turnover. Presently, serum or urinary assessments are used. However, the development of other procedures that are more patient-convenient, non-invasive and cost-efficient would significantly facilitate a clinician's ability to determine bone turnover. The objective of this application is to determine the feasibility of using saliva for this measurement. We will compare serum, urinary and salivary levels in 50 pre- and 50 post-menopausal women. Markers to be measured are bone alkaline phosphatase, osteocalcin, procollagen type propepties hydroxypyridinium crosslinks of collagen and crosslinked collagen telopeptides. Collection of saliva, serum and urine will be done at a single visit. We expect to observe reasonable good correlation between serum and saliva levels and poorer correlation between urine and saliva levels.

ELIGIBILITY:
Inclusion:

* 50 pre-menopausal females (25-40 yo)
* 50 post-menopausal females (55-70 yo)
* Good systemic health
* Good oral health

Exclusion:

* arthritis
* active periodontitis
* history or actively smoking
* diabetes
* HIV positive
* anti-coagulant therapy
* bone fracture within the past year
* pregnancy
* known metabolic bone disease

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subject population will be limited to pre-menopausal and post-menopausal females who are in good systemic health in an attempt to determine whether salivary levels of bone turnover markers hold valuable promise as a replacement or partner biofluid for serum and/or urine. In addition, proper selection of the subject population will minimize the effect of confounding variables. The specific inclusion criteria and exclusion criteria are listed below.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-05; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sreenivas Koka, D.D.S., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States